CLINICAL TRIAL: NCT02751476
Title: Effectiveness of Safe Drinking Water in Community Based Treatment of Severe Acute Malnutrition
Brief Title: Effectiveness of Safe Drinking Water in Treatment of Severe Acute Malnutrition (Pakistan)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Action Contre la Faim (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKG1A
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Marasmus
MeSH Terms: conditions — Protein-Energy Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- standard SAM treatment (control group) (Active Comparator): Standard Severe acute malnutrition treatment provided according to national nutrition protocol, in link with MoH health centers and structure.
  Interventions: Other: Standard Severe Acute Malnutrition Treatment
- SAM treatment + flocculent-disinfectant (Experimental): Standard Severe acute malnutrition treatment provided according to national nutrition protocol, in link with MoH health centers and structure. In addition, caregivers receive a flocculent-disinfectant for household level application.
  Interventions: Other: Point of Use (PoU) water treatment flocculent disinfectant.; Other: Standard Severe Acute Malnutrition Treatment
- SAM treatment + chlorine disinfectant (Experimental): Standard Severe acute malnutrition treatment provided according to national nutrition protocol, in link with MoH health centers and structure. In addition, caregivers receive a chlorine disinfectant for household level application.
  Interventions: Other: Point of Use (PoU) water treatment chlorine disinfectant; Other: Standard Severe Acute Malnutrition Treatment
- SAM treatment + ceramic water filter (Experimental): Standard Severe acute malnutrition treatment provided according to national nutrition protocol, in link with MoH health centers and structure. In addition, caregivers receive a ceramic water filter for household level application.
  Interventions: Device: Point of Use (PoU) ceramic water filter; Other: Standard Severe Acute Malnutrition Treatment

INTERVENTIONS:
Other: Point of Use (PoU) water treatment flocculent disinfectant. — A household level point of use water treatment of a flocculent disinfectant will be tested.
  Arms: SAM treatment + flocculent-disinfectant
Other: Point of Use (PoU) water treatment chlorine disinfectant — A household level point of use water treatment of a chlorine disinfectant will be tested.
  Arms: SAM treatment + chlorine disinfectant
Device: Point of Use (PoU) ceramic water filter — A household level point of use water treatment of a ceramic water filter will be tested.
  Arms: SAM treatment + ceramic water filter
Other: Standard Severe Acute Malnutrition Treatment — Standard CMAM treatment.

SUMMARY:
This study builds evidence on the importance of using safe drinking water during the nutritional treatment of children affected by Severe Acute Malnutrition (SAM). The following hypotheses will be tested: 1.The addition of safe drinking water to SAM treatment will reduce exposure to pathogens that cause diarrhoeal disease, thereby reducing diarrhoea incidence among enrolled children. 2.Reductions in pathogen exposure and diarrhoeal disease will result in shorter recovery pe-riods for children with SAM. The study will evaluate the effectiveness of safe drinking water in reducing SAM treatment cost and duration and will provide recommendations for improving SAM treatment protocols.

DETAILED DESCRIPTION:
A four group randomized control trial (RCT) will be used to evaluate the effectiveness of safe drinking water in SAM treatment protocols. Intervention groups will include: 1) standard SAM treatment (control group); 2) standard SAM treatment + flocculent-disinfectant water treatment (P&G Purifier of Water); 3) standard SAM treatment + chlorine disinfectant ("Aquatabs", a locally available mass market product); and 4) standard SAM treatment + ceramic water filter (locally available mass market product). All intervention groups will receive the standard SAM nutrition treatment and hygiene education. The control group will receive standard Community Managed Acute Malnutrition (CMAM) treatment only and households will use existing water treatment methods to represent the conventional CMAM program and to enable comparison with the other study arms (with improved water provision methods). A RCT was identified because it is a rigorous gold standard methodology design that is feasible given the context, and appropriate for determining whether or not safe drinking water is effective in CMAM programs. Site level randomization will be used and is preferable to individual randomization from a management perspective and because it increases likelihood of fidelity to the planned intervention. Limitations of the proposed design include 1) potential for bias because the study is not blinded and 2) possible contamination of the comparison groups. In order to minimize these risks, efforts will be made to geographically separate the comparison groups to reduce the risk of sharing of water treatment products. Blinding is not possible given the obviously different nature of the three PoU water treatment approaches and the need for a control group.

ELIGIBILITY:
Inclusion Criteria:

* Children in each selected community will be eligible for inclusion in the study if they are

  1. between six and 59 months of age,
  2. diagnosed as an uncomplicated SAM case
  3. enrolled in ACF's CMAMprogram
  4. if the child's caretaker gives consent for the child's participation.

Exclusion Criteria:

* Children will be ineligible for participation if

  1. they have a diagnosis of kwashiorkor; OR 2) they require in-patient treatment for SAM
  2. their caretakers are unwilling or unable to agree to their participation.
* Children graduating from in-patient treatment (i.e no remaining medical complications) to the out-patient CMAM program will be eligible for participation.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 820 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Recovery rate | 5 months
  the total number of cured children / total number of exited children (including cured, deceased, and lost to follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Doocy, PhD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Doocy S, Tappis H, Villeminot N, Suk A, Kumar D, Fazal S, Grant A, Pietzsch S. Point-of-use water treatment improves recovery rates among children with severe acute malnutrition in Pakistan: results from a site-randomized trial. Public Health Nutr. 2018 Nov;21(16):3080-3090. doi: 10.1017/S1368980018001647. Epub 2018 Aug 22. PMID 30132426